CLINICAL TRIAL: NCT04513405
Title: Role of Estrogens and Their Receptors in the Development of Skin Tears Evaluated in Residents of Residential Care Facilities.
Brief Title: Estrogens Levels and Receptors Status and Skin Tears
Acronym: ESKITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ER.CZ.2018.04
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Skin Tear; Estrogen Deficiency
Keywords: Skin Tears; Estrogen Receptors
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects with skin tears (Group A) (Other): A sample of peripheral venous blood will be taken to measure the levels of estrone and estradiol.
  A skin biopsy on the intact skin area near the skin tear will be performed.
  Interventions: Diagnostic Test: Blood sampling; Procedure: Shave Biopsy
- subjects without skin tears (Group B) (Other): A sample of peripheral venous blood will be taken to measure the levels of estrogen.
  A skin biopsy (thin layer) on the intact skin area of the arm will be performed in order to evaluate skin estrogen receptors.
  Interventions: Diagnostic Test: Blood sampling; Procedure: Shave Biopsy

INTERVENTIONS:
Diagnostic Test: Blood sampling — a peripheral venous blood sample will be analyzed to measure the levels of estrone and estradiol.
  The sample of the blood sample will be deposited in the red cap tube with a polymeric gel.
Procedure: Shave Biopsy — in the tissues, of the related estrogenic receptors, estrogen α receptors, estrogen β receptors (ER- α, ER-β) and G protein-coupled estrogen receptor 1 (GPER) correlates with the functional status of these receptors

SUMMARY:
Background: Skin tears (ST) or "laceration injuries" or "flap wounds" are injuries that are often found in residents of residential care facilities (RCFs). STs were first defined by Payne and Martin in 1993 as traumatic wounds, located mainly in the upper limbs, caused by "shearing, friction or mechanisms combined with the consequent separation of layers of skin. Skin Tears can cause psychological problems for the patient and represent an economic problem with important repercussions on both the patient and the community. The etiology suggests that the physiological changes of the skin related to old age, together with comorbidity, are among the main risk factors for their onset.

The precise data on the phenomenon are not many, but it is estimated that STs are much more frequent than the same pressure ulcers, observing prevalence rates in RCFs around 40% Therefore, there are several risk factors hypothesized so far. Much evidence has correlated, in various physiological or pathological conditions, the role of estrogens with the functions and aging of the skin.

Objectives: The project will develop on the analysis of populations of residents from RCFs belonging to the national territory. Two populations of residents cared in the RCF will be recruited. A group of subjects suffering from skin tears (group A) and a control group of subjects without skin tears (group B). The inclusion of patients in both groups will take place through a simple randomization procedure. Group A patients will be staged according to the STAR classification for skin tears. For each group a peripheral venous blood sample will be taken (to measure the levels of estrone and estradiol) and a skin biopsy will be performed in order to measure estrogen receptors (ERs) expression. A data collection sheet with angraphic and anamnestic data will be developed to correlate the demographic and comorbidity data with the clinical conditions of the patients and with the laboratory findings from the sampling.

Expected results: The primary endpoint will be the correlation between serum estrogen levels, receptor expression and the presence of skin tears. The secondary endopoint will be Correlation between receptor structure and clinical staging of skin tears.

Future prospectives: We believe that our study may open new frontiers in the prevention and in the management of these skin lesions.

DETAILED DESCRIPTION:
BACKGROUND Skin tears were firstly defined by Payne RL and Martin ML, and thereafter by more recent studies, as traumatic wounds occurring principally on the upper limbs, as a result of friction alone or shearing and friction forces, which separate the epidermis from the dermis (partial thickness wounds) or which separate both the epidermis and the dermis from underlying structures (full thickness wounds). Skin tears are reported to be a common wound especially on fragile exposed skin, which can be often encountered among older adult, disabled populations and neonates. Skin tears can be found on all areas of the body and are particularly common on the extremities. Skin tears may be also very common in public hospital (PH) inpatients and residents of residential care facilities (RCF) with prevalence up to 41% in these settings.

Skin Tears can cause psychological problems for the patient and represent an economic problem with important effects on both the patient and the community.

The risk factors hitherto hypothesized are many and include: advanced age, spasticity or rigidity, enticement, cognitive decline, long-term drug therapies, inadequate nutritional intake, etc but none of them, individually and independently, was found to be strongly correlated onset of skin tears, in such a way as to be able to effectively associate it with their onset.

Many evidences have correlated, in various physiological or pathological conditions, the role of estrogens with functions and skin aging.

The serum level of estrogens, and in particular estrone and estradiol, and the peripheral expression, in the tissues, of the related estrogenic receptors, estrogen α receptors, estrogen β receptors (ER- α, ER-β) and G protein-coupled estrogen receptor 1 (GPER) may be related to skin tears.

AIM The aim of the project is to study the correlation between serum estrogen levels and the expression of the related receptors, with the development of skin tears.

METHODOLOGY The project will develop on the analysis of populations of residents coming from ACF belonging to the national territory between a minimum of 10 and a maximum of 30. Each RCF will have to provide a number of subjects between 10 and 40.

The total patient sample will therefore be between a minimum of 100 and a maximum of 1200 subjects.

Therefore, two populations of guests assisted in the RCF will be recruited. A group of subjects affected by skin tears (group A) and a control group of subjects without skin tears (group B).

Patients will be included in both groups via a simple randomization procedure. The informed consent of the patient is required. A group of peripheral venous blood will be made to both groups to measure the levels of estrone and estradiol and a skin biopsy on the intact skin area near the lesion in group A and on a thin layer of healthy skin (Shave Biopsy) in the area of the arm in the control group (group B).

EXPECTED RESULTS Primary Endpoint The primary endpoint will be the correlation between serum estrogen levels, receptor expression and skin tears.

Secondary Endpoint. Correlation between receptorial structure and clinical staging of skin tears.

ELIGIBILITY:
Group A

Inclusion Criteria:

* Subjects of aged care facilities with skin tears

Exclusion Criteria:

* Patients who do not give consent;
* Inability of blood sampling and / or skin biopsy

Group B

Inclusion Criteria:

* Subjects of aged care facilities without skin tears

Exclusion Criteria:

* Patients who do not give consent;
* Inability of blood sampling and / or skin biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Estrogen and Skin Tears | at 1 year
  The primary outcome measure will be the correlation between serum estrogen levels and skin receptor expression and skin tears onset.

SECONDARY OUTCOMES:
Correlation between patient's estrogen status and clinical staging of skin tears | at 2 years
  The serum level of estrogens and the peripheral expression of estrogen receptor will be related to the severity of skin tears

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Study Chair — University Magna Graecia of Catanzaro; Nicola Ielapi, R.N., Principal Investigator — University La Sapienza of Rome
Locations (1):
- University La Sapienza of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payne RL, Martin ML. The epidemiology and management of skin tears in older adults. Ostomy Wound Manage. 1990 Jan-Feb;26:26-37. No abstract available. PMID 2306325
- [Background] Payne RL, Martin ML. Defining and classifying skin tears: need for a common language. Ostomy Wound Manage. 1993 Jun;39(5):16-20, 22-4, 26. PMID 8397703
- [Background] LeBlanc K, Baranoski S, Christensen D, Langemo D, Sammon MA, Edwards K, Holloway S, Gloeckner M, Williams A, Sibbald RG, Regan M. International Skin Tear Advisory Panel: a tool kit to aid in the prevention, assessment, and treatment of skin tears using a Simplified Classification System (c). Adv Skin Wound Care. 2013 Oct;26(10):459-76; quiz 477-8. doi: 10.1097/01.ASW.0000434056.04071.68. PMID 24045566
- [Background] El Safoury O, Rashid L, Ibrahim M. A study of androgen and estrogen receptors alpha, beta in skin tags. Indian J Dermatol. 2010;55(1):20-4. doi: 10.4103/0019-5154.60345. PMID 20418971
- [Background] Brincat MP, Baron YM, Galea R. Estrogens and the skin. Climacteric. 2005 Jun;8(2):110-23. doi: 10.1080/13697130500118100. PMID 16096167
- [Background] Serra R, Gallelli L, Perri P, De Francesco EM, Rigiracciolo DC, Mastroroberto P, Maggiolini M, de Franciscis S. Estrogen Receptors and Chronic Venous Disease. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):114-8. doi: 10.1016/j.ejvs.2016.04.020. Epub 2016 May 21. PMID 27220899
- [Background] Serra R, Ielapi N, Barbetta A, de Franciscis S. Skin tears and risk factors assessment: a systematic review on evidence-based medicine. Int Wound J. 2018 Feb;15(1):38-42. doi: 10.1111/iwj.12815. Epub 2017 Oct 17. PMID 29045078